CLINICAL TRIAL: NCT02010190
Title: Vascular Assessment in Adult Survivors of Childhood Cancer
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: VASCC
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Risk; Pediatric Cancer
Keywords: Pediatric malignancies; Cancer survivors; Coronary artery risk; Vascular function; Cardiovascular risk in survivors of pediatric cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer Survivors: Participants will be survivors of a childhood cancer.
- Control Group: Control participants will consist of age- and gender-matched individuals who are non-first-degree relatives of the survivor group.

SUMMARY:
This is an observational study that will collect data from adult survivors of childhood cancer and compare it to data collected from age- and gender-matched controls for the purpose of assessing vascular risk among cancer survivors.

Advances in cancer therapies have led to increasing numbers of adults previously treated for a pediatric malignancy, many of whom experience late adverse health-related sequelae and are at risk for developing chronic conditions related to their prior therapy. The epidemiology of many end-organ toxicities has been described, yet the pathophysiologic mechanisms of injury are incompletely understood. One mechanism may be damage to the circulatory system, in particular the endothelial layer, initiating an inflammatory state leading to dysfunction and premature atherosclerotic disease. This process may begin and significantly progress in a sub-clinical nature for many years prior to manifesting as a cardio- or cerebrovascular event. Using established and novel biomarkers predictive of atherosclerotic disease combined with unique measurements of vascular function, this study will assess pre-clinical vascular disease in a population of childhood and adolescent cancer survivors. The goals of this project are to investigate the effects of cancer therapy on the vascular system and acquire new knowledge with which to risk-stratify survivors and plan interventional studies to prevent or reduce premature vascular morbidity and mortality.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Evaluate biomarkers of vascular injury (inflammation, hemostasis, endothelial activation) among childhood cancer survivors compared to age/gender-matched controls.
* Assess vascular function among childhood cancer survivors compared to age/gender-matched controls.

SECONDARY OBJECTIVE:

* Investigate additional biomarkers of vascular health and function among childhood cancer survivors compared to age/gender-matched controls.

Eligible persons who consent to participate in this trial will be asked to do the following:

* Vital sign measurement including resting heart rate, blood pressure, height, and weight.
* Biomarker analysis will be completed by the Cytokine Reference Laboratory, Department of Pediatrics, University of Minnesota Medical School and the Vascular Biology Center (VBC), Department of Medicine, University of Minnesota Medical School.
* An echocardiogram to assess cardiac function.
* Pulse wave analysis will be measured with the CR-2000 Cardiovascular Profiling System.
* Pulse contour analysis will be studied using the Endo-PAT2000 system.
* Pulse wave velocity will be assessed using the SphygomoCor CVP Clinical System.

ELIGIBILITY:
INCLUSION CRITERIA:

* Cancer Survivors:

  * Treatment with chemotherapy and/or radiation therapy for a primary cancer diagnosed prior to age 21 years at St. Jude Children's Research Hospital (SJCRH).
  * ≥ 18 years of age at time of enrollment
  * Enrollment on the SJCRH SJLIFE protocol
  * No non-steroidal anti-inflammatory drug (NSAID) and/or aspirin (ASA) (≥ 325 mg) for 24 hours prior to testing.
* Control Group:

  * No history of or current treatment for any medical condition with therapeutic chemotherapy or radiation exposures
  * ≥18 years of age at time of enrollment
  * Enrolled on the SJCRH SJLIFE protocol as a community control
  * No NSAID and/or ASA (≥ 325 mg) for 24 hours prior to testing.

EXCLUSION CRITERIA:

* Active chronic inflammatory disease
* Diagnosis of sickle cell disease
* Current active infection
* On chronic anti-inflammatory medications
* History of upper extremity vascular bypass surgery or grafting.
* No active treatment with:

  * β- and α-adrenergic receptor antagonists (treat high blood pressure)
  * α-2 adrenergic agonists (treat high blood pressure)
  * Calcium channel antagonists (treat high blood pressure or chest pain)
  * HMG-CoA reductase inhibitors (treat high cholesterol)
  * Angiotensin-converting enzyme (ACE) inhibitors (treat high blood pressure, heart failure, and heart disease)
  * Angiotensin II receptor antagonists (treat high blood pressure and heart failure)
  * Diuretics (treat high blood pressure and heart failure)
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Currently pregnant (assessed by serum pregnancy test)
* A first-degree relative of a survivor participant (controls only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 202 potential cancer survivor participants will be recruited from the St. Jude Children's Research Hospital (SJCRH) SJLIFE Cohort Study and stratified by survival time (10-14, 15-19, 20-24, 25-29, and ≥ 30 years).
  202 potentially eligible comparison group participants will be recruited from the parent, sibling, relative or friend population who accompany patients to SJCRH. Control participants will not be a first-degree relative of a survivor participant. Potential comparison group members will be matched to potentially eligible participants by gender and age group.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean high sensitivity C-reactive protein (hsCRP) | Once, at first clinic visit
Mean fibrinogen | Once, at first clinic visit
Mean CEC surface expression of vascular cell adhesion molecule-1 (VCAM-1) | Once, at first clinic visit
Mean larger artery elasticity | Once, at first clinic visit

SECONDARY OUTCOMES:
Mean number of circulating endothelial cells (CECs) | Once, at first clinic visit
Mean CEC surface expression of P-selectin | Once, at first clinic visit
Mean soluble vascular cell adhesion molecule-1 (VCAM-1) | Once, at first clinic visit
Mean soluble P-selectin | Once, at first clinic visit
Mean von Willebrand factor (vWF) | Once, at first clinic visit
Mean D-dimer | Once, at first clinic visit
Mean plasminogen activator inhibitor-1 (PAI-1) | Once, at first clinic visit
Mean tissue-type plasminogen activator (tPA) | Once, at first clinic visit
Mean lipoprotein(a) | Once, at first clinic visit
Mean small artery elasticity (SAE) | Once, at first clinic visit
Mean reactive hyperemia peripheral arterial tonometry (RH-PAT) ratio | Once, at first clinic visit
Mean carotid-femoral pulse wave velocity | Once, at first clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Mulrooney, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols